CLINICAL TRIAL: NCT01475513
Title: Oral Contraceptives, Insulin Resistance and Cardiovascular Risk Profile in Pre-Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HM13769
Record Dates: First submitted 2011-11-08; First posted 2011-11-21 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Insulin Sensitivity; Cardiovascular Risk; Perimenopausal Disorder
Keywords: oral contraceptive; birth control pill; women; healthy volunteer; insulin sensitivity; insulin resistance; cardiovascular risk factors; endothelial function; estrogen metabolism; racial difference; glucose intolerance
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance | interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Same drug (orthocyclen) was administered to 2 groups (Caucasian women of reproductive age, and African American women of reproductive age)
Oversight: Data Monitoring Committee: No

ARMS (2):
- African-American women (Active Comparator): African-American women
  Interventions: Drug: Ortho Cyclen®
- Caucasian women (Active Comparator): Caucasian women
  Interventions: Drug: Ortho Cyclen®

INTERVENTIONS:
Drug: Ortho Cyclen® — Ethinyl estradiol 35 mcg and norgestimate 0.25 mg (oral) will be taken as one tablet daily for 21 days per month followed by a 7-day pill-free period per cycle. Duration of the study is for 6 cycles of this birth control pill.
  Other Names: Orthocyclen; Sprintec; Previfem; MonoNessa

SUMMARY:
Birth control pills are the most commonly used method of birth control. The purpose of this research study is to examine whether birth control pills change heart disease risk and how the body handles blood sugar when given to different women.

DETAILED DESCRIPTION:
The oral contraceptive pill is the most commonly used birth control method. It is debated whether the birth control pill affects how the body handles insulin and sugar, or whether the pill changes heart disease risk. The goal of this study is to evaluate whether certain factors, such as how the body processes hormones, and demographic factors (e.g. body weight and race), influence how the pill affects the handling of insulin and sugar, and heart health.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal, regular-cycling women 18-35 years
* Either African-American or Caucasian (African-American and Caucasian women will be BMI-matched)
* non-smoker.

Exclusion Criteria:

* Diabetes
* Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, and malignant disease
* Contraindications to oral contraceptive use (history of blood clots, heart attacks or stroke, vascular disease, coagulopathy, prolonged immobilization, breast cancer, migraine head-aches, major surgery within past 6 months, blood pressure >160/100 mmHg, pregnancy or lactation)
* Use of hormonal contraceptives, glucose-lowering medications, anti-hyperlipidemic, anti-hypertensive or other vasoactive drugs within previous 3 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05-28 (Actual); Study Completion 2014-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Cheang, Pharm. D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- African-American Women: African-American women
  Ortho Cyclen®: Ethinyl estradiol 35 mcg and norgestimate 0.25 mg (oral) took one tablet daily for 21 days per month followed by a 7-day pill-free period per cycle. Duration of the study is for 6 cycles of this birth control pill.
- Caucasian Women: Caucasian women
  Ortho Cyclen®: Ethinyl estradiol 35 mcg and norgestimate 0.25 mg (oral) took one tablet daily for 21 days per month followed by a 7-day pill-free period per cycle. Duration of the study is for 6 cycles of this birth control pill.
Period: Overall Study
Arm/Group | African-American Women | Caucasian Women
Started | 20 | 26
Completed | 17 | 16
Not Completed | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African-American Women | Caucasian Women | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.3 (3.43) | 21.6 (3.92) | 21.0 (3.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 0 | 18
  White | 0 | 17 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Sensitivity
Description: Insulin sensitivity from Frequently sampled IV glucose tolerance test (FSIVGTT), change from baseline to 6 months. Higher values indicate better insulin sensitivity
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: min ^ -1 / mIU / L
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 15
min ^ -1 / mIU / L | -1.91 [-5.63 to 1.80] | -5.63 [-9.47 to -1.80]

2. Primary Outcome: Change From Baseline in Flow-mediated Vasodilatation
Description: Change Flow-mediated Vasodilatation from baseline to 6 months. Higher values indicate less cardiovascular risk
Time Frame: Baseline, 6 months
Population: Data based on images. Some participants images could not be analyzed numerically.
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- African-American Women: African-American women
  Ortho Cyclen®: Ethinyl estradiol 35 mcg and norgestimate 0.25 mg (oral) was taken as one tablet daily for 21 days per month followed by a 7-day pill-free period per cycle. Duration of the study is for 6 cycles of this birth control pill.
- Caucasian Women: Caucasian women
  Ortho Cyclen®: Ethinyl estradiol 35 mcg and norgestimate 0.25 mg (oral) was taken as one tablet daily for 21 days per month followed by a 7-day pill-free period per cycle. Duration of the study is for 6 cycles of this birth control pill.
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 5 | 9
mm | 0.0503 [-0.0905 to 0.19099] | -0.0210 [-0.0868 to 0.04479]

3. Primary Outcome: Change From Baseline in Carotid Intima Media Thickness
Description: Change in Carotid Intima Media Thickness from baseline to 6 months, measured on the right carotid artery, posterior. Lower values indicate better cardiovascular risk profile
Time Frame: baseline, 6 months
Population: Data based on images. Some participants images could not be analyzed numerically.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 4 | 9
mm | -0.00008 [-0.0054 to 0.00523] | 0.00118 [-0.0024 to 0.00472]

4. Secondary Outcome: Change From Baseline in Acute Insulin Response to Glucose
Description: Acute Insulin Response to Glucose values obtained from FSIVGTT models--higher values indicate better insulin response
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mIU* L^-1 * min
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 17 | 15
mIU* L^-1 * min | -35.6 [-251.0 to 179.77] | 0.48 [-88.4 to 89.35]

5. Secondary Outcome: Change From Baseline in Glucose Effectiveness
Description: Obtained from FSIVGTT models--higher values indicate better effectiveness of glucose inducing its own disposition
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: 1000 * min ^ -1
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 15
1000 * min ^ -1 | -0.0255 [-0.0450 to -0.0059] | -0.0078 [-0.0134 to -0.0022]

6. Secondary Outcome: Change From Baseline in Disposition Index at 6 Months
Description: Modeled from FISVGTT--higher values indicate better glucose disposition
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: AIRG * Si
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 15
AIRG * Si | -911.73 [-2005 to 181.04] | -834.53 [-1963 to 294.09]

7. Secondary Outcome: Change From Baseline in Fasting Insulin at 6 Months
Description: Higher fasting insulin values indicate an increased metabolic risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: uIU/ mL
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 15 | 15
uIU/ mL | 1.66 [0.568 to 2.743] | 1.45 [0.363 to 2.537]

8. Secondary Outcome: Change From Baseline in Fasting Glucose at 6 Months
Description: Higher fasting glucose indicate an increased metabolic risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 15
mg/dL | -0.4 [-3.98 to 3.16] | 03 [-3.46 to 3.92]

9. Secondary Outcome: Change From Baseline in Areas-under-the-curve for Insulin at 6 Months
Description: Measured during oral glucose tolerance test. Higher values indicate increased metabolic risk
Time Frame: Baselines, 6 months
Measure: Mean (95% Confidence Interval); unit: mIU/mL * min
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 15 | 15
mIU/mL * min | 760.6 [-271.8 to 1733.1] | 1062.1 [29.7 to 2094.5]

10. Secondary Outcome: Change From Baseline in Areas-under-the-curve for Glucose
Description: Measured during oral glucose tolerance test. Higher values indicate increased metabolic risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL * min
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 15 | 15
mg/dL * min | 443.4 [-623.7 to 1510.4] | 514.2 [-552.8 to 1581.2]

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at 6 Months
Description: Higher value indicates increased cardiovascular risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 16
mmHg | 2.5 [-2.11 to 7.05] | -1.4 [-6.00 to 3.17]

12. Secondary Outcome: Change From Baseline in HDL at 6 Months
Description: Lower values indicate increased cardiovascular risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 16
mg/dL | 6.8 [3.69 to 9.94] | 6.9 [2.96 to 10.79]

13. Secondary Outcome: Change From Baseline in Body Mass Index in 6 Months
Description: Higher values indicate higher metabolic risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: Kg/m2
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 16
Kg/m2 | -0.32 [-0.886 to 0.253] | 0.39 [-0.669 to 1.456]

14. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to 6 Months
Description: Higher value indicates higher cardiovascular risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 16
mmHg | 0.6 [-2.64 to 3.89] | 2.44 [-0.83 to 5.70]

15. Secondary Outcome: Change in LDL From Baseline to 6 Months
Description: Higher value indicates higher cardiovascular risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 16
mg/dL | 13.4 [5.71 to 21.04] | 17.1 [6.10 to 28.15]

16. Secondary Outcome: Change in Triglycerides From Baseline to 6 Months
Description: Higher values indicate higher cardiovascular risk
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | African-American Women | Caucasian Women
Number analyzed (Participants) | 16 | 16
mg/dL | 13.3 [-3.78 to 30.28] | 29.3 [4.23 to 54.27]

ADVERSE EVENTS:
Time Frame: Post-baseline follow-up phone call at 10 days
Description: Superficial venous thrombosis at IV site
Arm/Group | African-American Women | Caucasian Women
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/26
Other Adverse Events (participants affected / at risk) | 0/20 | 0/26

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed. Some subjects did not have reportable carotid intima media thickness and flow mediated dilatation values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes